CLINICAL TRIAL: NCT07099625
Title: Optimization of Adaptive Rowing Seating (OARS)
Brief Title: Optimization of Adaptive Rowing Seating
Acronym: OARS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Louis Stokes VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RRD5-015-24W
Record Dates: First submitted 2025-07-07; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Diseases; Spinal Cord Injuries; Neurodegenerative Disorders; Cerebrovascular Accident With Associated Sequelae
Keywords: Veteran Health; Sports for Persons with Disabilities; Paralysis; Paresis; Adaptive Sports; Indoor Rowing
MeSH Terms: conditions — Spinal Cord Diseases; Spinal Cord Injuries; Neurodegenerative Diseases; Paralysis; Paresis

STUDY DESIGN:
Intervention Model Description: Single group assignment with crossover design where participants will be randomized which rowing seat they start with and which seat is second. n=15
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- AIRS V2 (Experimental): The (Adaptive Indoor Rowing Seat) AIRS V2 will be used within an established adaptive rowing protocol for Veterans with limited trunk strength and compared with the Paddle Sport adaptive seating system.
  Interventions: Device: Adaptive Indoor Rowing Seat
- Paddle Sport Adaptive Seating System (Experimental): The (Adaptive Indoor Rowing Seat) AIRS V2 will be used within an established adaptive rowing protocol for Veterans with limited trunk strength and compared with the Paddle Sport adaptive seating system.
  Interventions: Device: Paddle Sport adaptive seating system

INTERVENTIONS:
Device: Adaptive Indoor Rowing Seat — Light weight adjustable indoor rowing seat for Veterans with limited trunk stability.
  Other Names: AIRS V2
  Arms: AIRS V2
Device: Paddle Sport adaptive seating system — On market comparator (discontinued) adaptive indoor rowing seat for individuals with limited trunk stability.
  Arms: Paddle Sport Adaptive Seating System

SUMMARY:
Adaptive sports programs are integral components to combating Veteran isolation, promoting wellbeing and seeking to build teams, networks, communities. These activity-based communities are medicine free treatment systems enhancing Veterans' health from a holistic perspective. This approach to Veteran healthcare is critical as studies indicate Veterans not only have 56% higher perceived social isolation but are also 1.5x more susceptible to suicide than the general public. It is imperative to improve access to exercise and physical activity through adaptive sport or recreation. This proposal is going to focus on Adaptive Indoor Rowing for Veterans with limited or changing trunk stability (i.e. SCI/D, paralysis, paresis, etc.). Rowing is a unique full-body activity that increases cardiovascular demand and increases coordination and aerobic capacity through movement. This proposal aims to address critical gaps in adaptive rowing technology and provide Veterans with limited trunk stability access to full stroke adaptive rowing.

DETAILED DESCRIPTION:
Significance to VA: Veterans with SCI/D experience limited access to physical activity due to insufficient adaptive equipment options. It is imperative to improve access to exercise and physical activity through the thoughtful design and development of adequate adaptive technologies that reduce barriers to participation. The current state of adaptive indoor rowing is ineffective at exercising the full body, which limits the improvement of cardiovascular health and neuromusculoskeletal coordination resulting in decreased benefits to Veterans and may discourage further motivation to participate. This proposal focuses on Adaptive Rowing for Veterans with limited trunk stability and specifically on the need for new adaptive seat options for indoor rowing

Innovation and Impact: Current adaptations for indoor rowing bypass the use of the legs and reduce participant range of motion, limiting the full-body exercise to an arms-only workout regardless of the user's ability. The proposed adaptive indoor rowing seat provides a full slide motion while also regulating trunk range of motion movements. A function that is currently unavailable in any current or past adaptive indoor rowing seat.

Specific Aims:

1) Optimize a new clinically viable adaptive indoor rowing seat for Veterans with limited trunk stability.

Subtask 1) Assess 1st prototype of Adaptive Indoor Rowing Seat (AIRS V1) with Veterans and clinicians specializing in SCI/D and collect feedback.

Subtask 2) Develop 2nd prototype of Adaptive Indoor Rowing Seat (AIRS V2) from Veteran and clinician feedback collected in Subtask 1.

Subtask 3) Test feasibility of 2nd prototype of Adaptive Indoor Rowing Seat (AIRS V2) with Veterans in Cleveland and collect feedback from Veterans and clinicians.

H1) The AIRS V2 will result in increased anterior/posterior trunk movement when compared to the discontinued Paddle Sport adaptive seating system while performing rowing.

H2) Rowing with the AIRS V2 will result in increased stroke length or ability to generate more power through their upper extremities when compared to the discontinued Paddle Sport adaptive seating system.

H3) Veterans will rate feeling more stable and comfortable rowing with the AIRS V2.

Subtask 4) Generate 3rd prototype (AIRS V3) from feedback on AIRS V2. The entirety of feedback collected, and data analyzed will result in the development of two AIRS V3 prototypes.

Methodology: Year one of this proposal will focus on Subtask 1 and 2. First, feedback on the design of AIRS V1 will be collected from Veterans with SCI/D and SCI/D Clinicians at the 2025 National Wheelchair Games being hosted in Minneapolis and the RECOVER and APT Center Veteran Engagement Panels. Feedback will also be obtained from study industry partners: Concept2 and US Rowing. The investigators will then design and fabricate AIRS V2 incorporating the Veterans with SCI/D, SCI/D clinicians, and industry feedback. In year 2, AIRS V2 will be shipped to the APT Center for human subject testing with Veterans with SCI/D. The hypotheses listed above will be tested to access whether AIRS V2 is more effective and preferred than the Paddle Sport adaptive seating system currently being used at the APT Center: Both sites will work together to use the data and feedback from the human subjects testing to guide any additional modifications needed for AIRS V3. In Year 3, the design team will build two AIRS V3s, shipping one to the APT Center, as well as disseminating any remaining findings.

Path to Translation/Implementation: Additionally, the overall experience and insights gained throughout this project will contribute to commercialization opportunities of AIRS V3. Throughout this proposal the investigators will strategize with study industry partners, Concept2 & US Rowing, along with VA Technology Transfer Program to determine the best commercialization path for getting the AIRS V3 in the hands of Veterans.

ELIGIBILITY:
Inclusion Criteria:

* Non-ventilator dependent paralysis, such as:

  * central nervous system impairment
  * spinal cord injuries with single neurological level in the cervical to lumbosacral region
  * cerebrovascular accident with associated sequelae including but not limited to hemiparesis and spasticity
  * neurodegenerative disorders including but not limited to amyotrophic lateral sclerosis, multiple sclerosis, multiple system atrophy, and parkinsonism
* Poor trunk control/stability
* Ability of body structure to fit within the limits of AIRS and the rowing system
* Either volitional control of lower extremities or response/tolerance to electrical stimulation
* Individuals who would be classified as PR2 or PR1 - FISA Para-Rowing Classifications

Exclusion Criteria:

* Veterans will be excluded if they have:

  * acute illness or injury
  * active or recent pressure injuries in the last 6 months affecting their ability to safely row (e.g., the coccyx, ischial tuberosity, sacrum, etc.)
* Individuals who would be classified as NE or PR3-PD - FISA Para-Rowing Classifications
* Flap procedure to address pressure injury less than one year prior
* Upper extremity pain that restricts rowing
* Surgical procedure within past 6 months that would make the study procedures unsafe (e.g., tendon repairs/transfers, neural decompressions, bony fusions, etc.)
* Upper extremity or spine fractures within past 3 months, or longer if remains unstable/not fully healed.
* Medical conditions such as cardiovascular disease, pulmonary disease, or other conditions that would make the study procedures unsafe pregnancy
* Inability to communicate with the study team in real time
* Inability to follow simple commands
* Unable or unwilling to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-07-06 (Estimated); Primary Completion 2027-07-05 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Trunk Movement | up to 4 weeks after enrollment
  Changes in angular trunk position (degrees) will be captured during a self-selected, moderate pace for 2-5 minutes depending on their ability. They will complete 3 trials of rowing with at least 10 minutes of rest between trials on each seat.
Rowing Stroke Length | up to 4 weeks after enrollment
  Changes in stroke length (cm) will be captured during a self-selected, moderate pace for 2-5 minutes depending on their ability. They will complete 3 trials of rowing with at least 10 minutes of rest between trials on each seat.
Power (Watts) | up to 4 weeks after enrollment
  Changes in power generation (Watts) will be captured during a self-selected, moderate pace for 2-5 minutes depending on their ability. They will complete 3 trials of rowing with at least 10 minutes of rest between trials on each seat.
Custom Usability Items | up to 4 weeks after enrollment
  Questions study specific to the usability of the indoor rowing seats
System Usability Score (SUS) [Brook (1996, 2013)] | up to 4 weeks after enrollment
  Widely used measure to assess usability of any technological system. It is a questionnaire based approach that combines subjective ratings and objective metrics to provide a quantitative measure of usability.
User Experience Questionnaire (UEQ) [(Laugwitz et al 2006, 2008)] | up to 4 weeks after enrollment
  A quick and comprehensive assessment tool that allows users "in a very simple and immediate way to express feelings, impressions, and attitudes that arise when experiencing the product under investigation."
Usability Metric for User Experience [(Finstad et al 2010)] | up to 4 weeks after enrollment
  Usability experience survey

CONTACTS AND LOCATIONS:
Overall Officials: John M Looft, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (2):
- United States (2):
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota
  - Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No